CLINICAL TRIAL: NCT03539354
Title: TEmporary Spinal CoRd StiMulatIon to PrevenNt Atrial FibrillaTION AFter Cardiac Surgery (TerminationAF)
Brief Title: TEmporary Spinal CoRd StiMulatIon to PrevenNt Atrial FibrillaTION AFter Cardiac Surgery
Acronym: TerminationAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TERMAF1
Record Dates: First submitted 2018-04-23; First posted 2018-05-29 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation
Keywords: Atrial fibrillation; Spinal cord stimulatoin; Coronary artery bypass grafting
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation | interventions — Coronary Artery Bypass; Endothelin B Receptor Antagonists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CABG + b-blockers (Active Comparator): Standart coronary artery bypass grafting is performed with b-blockers treatment. Continuous ECG during intensive care unit stay, daily ECG, and 24-h Holter monitor recordings will be performed at 7, 14, 21, and 30 days after coronary artery bypass grafting, external loop recorder after discharge from intensive care unit till 30 days after coronary artery bypass grafting.
  Interventions: Procedure: Coronary artery bypass grafting; Drug: B-blockers
- CABG + b-blockers + temporary SCS (Experimental): Before coronary artery bypass grafting in the experimental group, 3 days of temporary spinal cord stimulation is performed than device turned off and coronary artery bypass grafting procedure is made. The device for spinal cord is turned on in intensive care unit for 7 days. Continuous ECG during intensive care unit stay, daily ECG, and 24-h Holter monitor recordings will be performed at 7, 14, 21, and 30 days after coronary artery bypass grafting, external loop recorder after discharge from intensive care unit till 30 days after coronary artery bypass grafting.
  Interventions: Device: Temporary spinal cord stimulation; Procedure: Coronary artery bypass grafting; Drug: B-blockers

INTERVENTIONS:
Device: Temporary spinal cord stimulation — Percutaneous trial (temporary) electrodes are placed through a 14-gauge needle.The skin is entered at the medial aspect of the pedicle with the Tuohy needle usually angled 30-45° toward the midline for optimal entry into the epidural space at the interlaminar edge 1 or 2 levels of cephalad (usually, Th5-Th6 level). The 14-gauge needle is then passed with the bevel facing up at a 30-45° oblique angle to reach the depth of the midline laminar target.The Tuohy needle is then carefully removed and the operative site is cleaned with chlorhexidine and alcohol. Temporary stimulation is carried out till coronary artery bypass grafting surgery for 3 days, then stimulation turns off during surgery. At the end of coronary artery bypass grafting the temporary stimulation turns on in the intensive care unit and continues for 7 days. After that, the temporary leads will be removed.
  Arms: CABG + b-blockers + temporary SCS
Procedure: Coronary artery bypass grafting — Standart coronary artery bypass grafting procedure.
Drug: B-blockers — Standart b-blocker therapy will be administered in each group for AF prophylactics

SUMMARY:
To compare of atrial arrhythmia incidence in patients with coronary artery disease and atrial fibrillation history, undergoing either coronary artery bypass grafting plus temporary spinal cord stimulation or coronary artery bypass grafting alone

DETAILED DESCRIPTION:
The study includes 60 patients. Patients are randomized into 2 groups: coronary artery bypass grafting plus b-blocker treatment (according to guidelines; group I) and coronary artery bypass grafting plus b-blocker treatment (according to guidelines) plus temporary spinal cord stimulation (group 2). Temporary spinal cord stimulation is performed for 3 days before surgery and 7 days after coronary artery bypass grafting. Continuous ECG during intensive care unit stay, daily ECG and 24-h Holter monitor recordings at 7, 14, 21, and 30 days after coronary artery bypass grafting, external loop recorder after discharge from intensive care unit until 30 days after coronary artery bypass grafting. Rhythm status and clinical outcome assessment at 12 month follow up

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years;
* indications for coronary artery bypass grafting according to guidelines;
* pre-operative history of paroxysmal atrial fibrillation;
* absent of contraindications for spinal cord stimulation;
* signed inform consent.

Exclusion Criteria:

* previous heart surgery or atrial fibrillation ablation procedure;
* emergency coronary artery bypass grafting;
* left ventricle ejection fraction <35%;
* unstable angina or heart failure;
* persistent atrial fibrillation or atrial fibrillation at the time of screening;
* planned Maze procedure or pulmonary vein isolation;
* use of class I or III antiarrhythmic drugs within 5 elimination half-lives of the drug;
* need for concomitant valve surgery;
* Inability to control the device for spinal cord stimulation;
* coagulopathy, immunosuppression, or other condition associated with an unacceptable surgical risk for spinal cord stimulation;
* Need for therapeutic diathermy in the area of leads placement;
* Need for pacemaker/ICD/CRT-D implantation;
* unwillingness to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events | 30 days
  MACE (Death, Stroke/TIA, Myocardial infarction), acute kidney injury, spinal cord injury
Occurrence of atrial tachyarrhythmias | 30 days
  Occurrence of any atrial tachyarrhythmias including atrial fibrillation, atrial tachycardia, atrial flutter lasting ≥ 30 sec during 30 days after surgery
Occurrence of tachyarrhythmias | 12 months
  Occurrence of any atrial tachyarrhythmias including atrial fibrillation, atrial tachycardia, atrial flutter lasting ≥ 30 sec 30 days after surgery

SECONDARY OUTCOMES:
Marker of myocardial injury - high-sensitive Troponin I | 30 days
Marker of myocardial injury - CK-MB | 30 days
Marker of kidney injury - Creatinine | 30 days
Hemodynamic parameter - Blood pressure | 30 days
  Invasive blood pressure, pulmonary artery pressure, central venous pressure, pulmonary artery wedge pressure
Hemodynamic parameter - Heart rate | 30 days
Hemodynamic parameter - Cardiac index | 30 days
Hemodynamic parameter - Vascular resistance | 30 days
  Systemic vascular resistance, pulmonary artery resistance
Acute pain assessment | 30 days
  The Wong-Baker Faces Pain Rating Scale
Inotropic score | 30 days
Duration of mechanical ventilation | 30 days
Duration of intensive care unit stay | 30 days
Renal-replacement therapy | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - MedElect Clinic, Moscow
  - Novosibirsk Research Institute of Circulation Pathology, Novosibirsk

REFERENCES:
- [Derived] Romanov A, Lomivorotov V, Chernyavskiy A, Murtazin V, Kliver E, Ponomarev D, Mikheenko I, Yakovlev A, Yakovleva M, Steinberg JS. Temporary Spinal Cord Stimulation to Prevent Postcardiac Surgery Atrial Fibrillation: 30-Day Safety and Efficacy Outcomes. J Am Coll Cardiol. 2022 Feb 22;79(7):754-756. doi: 10.1016/j.jacc.2021.08.078. No abstract available. PMID 35177200